CLINICAL TRIAL: NCT04322084
Title: Continuous Ambulatory Monitoring to Predict Elevated Risk of Infection in Children With Lymphoblastic Leukemia Undergoing Induction Chemotherapy (CAMPER-ALL)
Status: Withdrawn | Type: Observational
Why Stopped: The study was activated at the onset of the COVID pandemic. At that time voluntary, non-therapeutic research was placed on hold. Now the technology has evolved and have elected to forego this protocol.
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CAMPER-ALL; NCI-2011-01222 (Registry Identifier: NCI)
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Participants: Participants will be enrolled during induction therapy for ALL, before the first high-risk period of treatment, and will contribute data for two 5-day periods of continuous monitoring.
  Interventions: Other: Wearable Sensors

INTERVENTIONS:
Other: Wearable Sensors — To develop predictive algorithms that identify early onset of sepsis in children being treated for ALL. This study will use a two-stage design. The initial stage (the feasibility phase) will evaluate the feasibility of data collection, and the second stage (the completion phase) will provide data for the design of predictive models.

SUMMARY:
Acute lymphoblastic leukemia (ALL) is the most common cancer of childhood and long-term survival has risen to above 90%, but 1-4% of treated patients die from infections. Early detection and treatment of infection can improve these outcomes by preventing increased severity and death. This study aims to determine whether continuous analysis of information from wearable devices (Like a watch and sticky patch) that measure temperature, pulse rate, oxygen level, and other similar information can predict infection before it is apparent to the patient or caregiver. About 65 patients will be enrolled and will wear these devices for 10 days; during that time the information will be recorded, but not available. After completion, information collected immediately before infection will be compared to other times to identify features that predict infections.

DETAILED DESCRIPTION:
Primary Objectives (Feasibility Phase) To determine the feasibility of non-invasive collection of continuous physiological data in children with acute lymphoblastic leukemia during outpatient treatment.

(Completion Phase) To develop competing sepsis prediction algorithms using continuous physiological data during outpatient treatment in children with acute lymphoblastic leukemia during high-risk periods of induction therapy.

Secondary Objectives To estimate the PPV and NPV of competing sepsis prediction algorithms using continuous physiological data for prediction of fever and sepsis in children with acute lymphoblastic leukemia during high-risk periods of induction therapy.

To estimate the frequency of undocumented fever episodes in children with acute lymphoblastic leukemia during high-risk periods of induction therapy.

To estimate the time from detection of fever or sepsis by a wearable device to identification by standard practice in children with acute lymphoblastic leukemia during high-risk periods of induction therapy.

This study aims to determine whether continuous analysis of those biosignals in children treated for ALL can predict early onset of sepsis. To collect those biosignals, we combine two wearable sensors, namely TempTraq, an adhesive temperature sensor, and Empatica E4, a wearable physiological monitoring device.

Data will be collected during two selected high-risk 5-day periods of induction therapy for acute lymphoblastic leukemia. Statistical models will be applied and a series of validation methodologies will be developed to arrive at an optimal predictive model for subsequent external validation .

This study will use a two-stage design. The initial stage (the feasibility phase) will evaluate the feasibility of data collection, and the second stage (the completion phase) will provide sufficient data for the development of predictive models and the estimation of the sensitivity and specificity of these models .

Feasibility Phase

The feasibility phase of the study will comprise the first 10 study participants, including at least 3 in each age group (5 to <10 years, and >/= 10 years). The aim of this stage is to estimate the proportion of time that continuous monitoring data are available, and these results will determine whether the study progresses to the completion phase

Completion Phase

The Completion Phase will comprise approximately 55 participants. Enrollment will continue until:

1. A total of 15 participants have experienced a fever or sepsis event for the prediction model, and
2. At least 15 participants have completed the study without experiencing a fever or sepsis event.

ELIGIBILITY:
Inclusion Criteria:

* Between 5 and 25 years of age at time of study enrollment
* Undergoing induction therapy for acute lymphoblastic leukemia at St. Jude
* Expected to remain outpatient during periods of high infection risk

Exclusion Criteria:

* Documented allergy to components of the device (Empatica E4: elemental silver, polyurethane, or polycarbonate; TempTraq: latex-free adhesive).
* Any condition that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol
* Current fever or sepsis at time of enrollment

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All Participants who meet eligibility criteria and consent to enrollment on the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility phase | 5 weeks
  The aim of this stage is to estimate the proportion of time that continuous monitoring data are available, and these results will determine whether the study progresses to the completion phase.
Completion phase | 5 weeks
  This phase will provide sufficient data to develop competing sepsis prediction algorithms using continuous physiologic data for cross-validation.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Wolf, MBBS, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: clinical Trials Open at St. Jude — http://www.stjude.org/protocols